CLINICAL TRIAL: NCT03936504
Title: Clinical Efficacy and Mechanism of Tai Chi Cardiac Rehabilitation Program（TCCRP） in Patients With Chronic Coronary Syndrome Under Fusion Cardiac Rehabilitation Model: a Randomized Controlled Trial
Brief Title: Efficacy and Mechanism of TCCRP in Patients With Chronic Coronary Syndrome Under Fusion Cardiac Rehabilitation Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Normal University (Other)
Responsible Party: Principal Investigator, Jing Ma, Clincial professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S2019-060-03
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Coronary Heart Disease; Chronic Coronary Syndrome
Keywords: Tai Chi; Cardiac rehabilitation; Chronic coronary syndrome; Safety; Effectiveness; Randomized controlled trial; Fusion cardiac rehabilitation model
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Group received conventional exercise rehabilitation programs (CERP).
  Interventions: Behavioral: Control Group ：conventional exercise rehabilitation programs (CERP)
- Experimental Group (Experimental): Group received Tai Chi cardiac rehabilitation program(TCCRP).
  Interventions: Behavioral: Experimental Group ：Tai Chi cardiac rehabilitation program (TCCRP)

INTERVENTIONS:
Behavioral: Control Group ：conventional exercise rehabilitation programs (CERP) — The participants in the control group will receive a conventional exercise rehabilitation programs (CERP) thrice a week for 12 weeks. Each training session lasts for 60 minutes, including ordinary warm-up exercises (10 minutes), aerobic activity (30 minutes), resistive exercise (10 minutes), and cool-down exercises(10 minutes). Each training session includes:(1) an active warm-up including arm-swinging, gentle stretches of the neck, shoulders, spine, arms, legs and so on;(2) aerobic activity mainly including aerobic radio exercise;(3) resistive exercise mainly including elastic belt exercise;(4) cool-down session involving active and static stretching exercises with primary body movements.
  Arms: Control Group
Behavioral: Experimental Group ：Tai Chi cardiac rehabilitation program (TCCRP) — Participants perform Tai Chi cardiac rehabilitation program(TCCRP) thrice a week for 12 weeks. Each training session lasts for 60 minutes, including Tai Chi warm-up exercises(10 minutes), Bafa Wubu of Tai Chi(30 minutes), Tai-Chi in conjunction with X-light-band resistance exercise(10 minutes), and Tai Chi cool-down exercises(10 minutes). All participants are encouraged to practice Tai Chi followed the instructional video until finishing 12-week exercise.
  Arms: Experimental Group

SUMMARY:
This study is a prospective, multi-center, randomized controlled clinical study. It developed an innovative Tai Chi Cardiac Rehabilitation Program (TCCRP) for patients with chronic coronary syndrome (CCS) and evaluated the efficacy, acceptability and safety of TCCRP on patients with CCS in order to explore the possible mechanism of its feasibility.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled clinical trial of 100 participants with chronic coronary syndrome (CCS) that compares Tai Chi cardiac rehabilitation program (TCCRP) with conventional exercise rehabilitation programs (CERP), with an allocation ratio of 1:1. A total of 6 months study period, including 1 month in-hospital rehabilitation, 2 months home-based rehabilitation and 3 months follow-up. The main outcome indicators were measured at baseline, 1 month, 3 months and 6 months. The secondary outcome measures will be measured at baseline and at 3 months.

ELIGIBILITY:
Inclusion criteria

1. Male or non-pregnant women aged from 18 to 80 years;
2. Patients who met the stable angina pectoris in accordance with coronary heart disease;
3. NYHA class Ι, Π or Ш;
4. Participants were able to understand the purpose of clinical trials and voluntarily participate and sign informed consent.

Exclusion criteria

1. Acute myocardial infarction (AMI) within 2 weeks;
2. Severe aortic stenosis;
3. Hypertrophic cardiomyopathy;
4. Severe valvular heart disease;
5. Malignant tachyarrhythmia;
6. The patient compliance was poor and the clinical trial could not be completed according to the requirements.
7. Combined exercise can cause deterioration of the nervous system, motor system disease, or rheumatic disease.
8. In the past 3 months, those who regularly practice Tai Chi;
9. Patients with gastrointestinal diseases, infectious diseases, renal insufficiency, and a history of gastrointestinal surgery within one year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in score of Chinese Perceived Stress Scale (CPSS) | baseline, 1 month, 3 months, 6 months
  Chinese Perceived Stress Scale is a self-rated questionnaire, which assesses perceived stress. Chinese Perceived Stress Scale is consisted of 14 items, which are divided into two dimensions: sense of tension and loss of control. Higher scores indicate higher levels of stress，lower scores indicate lower levels of stress. Chinese Perceived Stress Scale will be evaluated at baseline, 1 month, 3 months and 6 months.
Change in score of Medical Outcomes Study Questionnaire Short Form 36 Health Survey (36-Item Short Form Survey) | baseline,1 month, 3 months, 6 months
  SF-36 Health Survey(SF-36) . This is a multi-purpose, short-form health survey with only 36 questions. SF-36 items cover eight domains: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. Higher scores indicate higher levels of health. SF-36 will be evaluated at baseline, 1 month, 3 months and 6 months.
6-minute walk test (6 MWT) | baseline, 1 month, 3 months, 6months
  6-minute walk test (6 MWT). 6MWT measures the distance a patient can walk quickly on a flat, hard ground in 6 minutes. 6MWT will be evaluated at baseline, 1 month, 3 months and 6 months.

SECONDARY OUTCOMES:
Body fat rate | baseline, 3 months
  Body fat rate will be tested by the Inbody770 at baseline and 3 months (at the end of the intervention) through bioelectrical impedance analysis.
Peak oxygen uptake（VO2Peak） | baseline, 3 months
  Cardiopulmonary exercise test (CPET) is an objective method being increasingly used in a wide spectrum of clinical practice for assessing the functional capacity of patient with coronary heart disease. Peak oxygen uptake（VO2Peak）will be tested by CPET at baseline and 3 months (at the end of the intervention).
Locomotor skills | baseline，3 months
  Locomotor skills includes handgrip strength, balance and flexibility. Handgrip strength, which is used to determine the maximum isometric strength of the hand and forearm muscles, will be measured using the handgrip strength dynamometer produced by CAMRY (product type EH101). The best result from repeated tests of each hand will be recorded. The balance test mainly includes standing on one foot with eyes closed, standing on one foot with eyes open, standing in situ with closed eyes and so on. Flexibility will be measured by seated forward flexion test. Locomotor skills will be evaluated at baseline and at the end of the 3-month intervention.
Left ventricular ejection fraction(LVEF) | baseline, 3 months
  LVED Vi and LVEF are also to be assessed using echocardiography at baseline and at the end of the 12-week intervention.
Heart rate variability | baseline, 3 months
  Heart rate variability will be assessed at baseline and at the end of the 3-month intervention.
Low-density lipoprotein | baseline, 3 months
  Low-density lipoprotein inspections will be tested at baseline and at the end of the 3-month intervention using an automatic biochemical analyzer.
Testing of intestinal flora | baseline, 3 months
  Intestinal flora tests will be evaluated at baseline and at the end of the 3-month intervention.

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | baseline, 3 months
  Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report measure. The GAD-7 asks how often participants have been bothered by anxiety symptoms in the past 2 weeks. Items are rated on a 4-point Likert scale indicating symptom frequency, ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with higher scores indicating GAD. According to the original authors, the total score can then be interpreted as indicating no/minimal anxiety (0-4), mild (5-9), moderate (10-14), or severe (15-21), with a reasonable cut-off value for identifying cases of GAD at 10 points. GAD-7 will be evaluated at baseline and at the end of the 3-month intervention.
Patient Health Questionnaire-9 (PHQ-9) | baseline, 3 months
  The Patient Health Questionnaire-9 (PHQ-9) is designed for use with adults in assessing and monitoring depression severity based on Diagnostic and Statistical Manual of Mental Disorders (4th ed.;DSM-IV); The PHQ-9 asks clients to check off the number of days they have been bothered by each of the PHQ-9 symptoms over the"last two weeks." The nine items, based on DSM criteria for diagnosis of depression, are used to generate scores of 0, 1, 2, or 3 to the response categories of "not at all," "several days," "more than half the days," and "nearly every day,". The higher the score, the more serious the depression. PHQ-9 will be evaluated at baseline and at the end of the 3-month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, doctor, Principal Investigator — Department of Cardiology in Chinese PLA General Hospital
Locations (3):
- China (3):
  - Beijing Water Conservancy Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chaoyang District Anzhen Community Health Service Center, Beijing

IPD SHARING:
Plan to Share IPD: Yes
6 months after republication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The IPD of the publication will be shared, including characteristic data,results, clinical follow up data.

REFERENCES:
- [Background] Yang YL, Wang YH, Wang SR, Shi PS, Wang C. The Effect of Tai Chi on Cardiorespiratory Fitness for Coronary Disease Rehabilitation: A Systematic Review and Meta-Analysis. Front Physiol. 2018 Jan 4;8:1091. doi: 10.3389/fphys.2017.01091. eCollection 2017. PMID 29354065
- [Background] Pozzan R, Da Cruz P di M, Castier MB, Barbosa EC, Barbosa JS, Da Rocha PJ, Albanesi Filho FM, Ginefra P, Gomes Filho JB. [Cardiac rehabilitation of patients with coronary disease. Evaluation after 3 and 6 months of aerobic training at the community level]. Arq Bras Cardiol. 1988 May;50(5):305-10. No abstract available. Portuguese. PMID 3240110
- [Background] Ferguson RJ, Bourassa MG, Cote P, Chaitman BR. [Cardiovascular effects of exercise and physical training in coronary disease]. Union Med Can. 1979 Oct;108(10):1187-94. No abstract available. French. PMID 392869
- [Background] Fernandes F, Morais C, Esteves M, Camilo V, Nazare J, da Cunha JC, Amram SS. [Atrial pacing and the exercise test in the evaluation of coronary disease. A comparative study]. Rev Port Cardiol. 1990 Sep;9(9):675-9. Portuguese. PMID 2257154
- [Background] Hartung GH. Diet and exercise in the regulation of plasma lipids and lipoproteins in patients at risk of coronary disease. Sports Med. 1984 Nov-Dec;1(6):413-8. doi: 10.2165/00007256-198401060-00001. No abstract available. PMID 6390610
- [Background] Ferguson RJ, Petitclerc R, Choquette G, Chaniotis L, Gauthier P, Huot R, Allard C, Jankowski L, Campeau L. Effect of physical training on treadmill exercise capacity, collateral circulation and progression of coronary disease. Am J Cardiol. 1974 Dec;34(7):764-9. doi: 10.1016/0002-9149(74)90693-6. No abstract available. PMID 4432806
- [Background] Lepretre PM, Ghannem M, Bulvestre M, Ahmaidi S, Delanaud S, Weissland T, Lopes P. Exercise-based Cardiac Rehabilitation in Coronary Disease: Training Impulse or Modalities? Int J Sports Med. 2016 Dec;37(14):1144-1149. doi: 10.1055/s-0042-112591. Epub 2016 Nov 10. PMID 27832671
- [Background] Sharma S, Malhotra A. Exercise testing and coronary disease: pushing fitness to higher peaks. Eur Heart J. 2019 May 21;40(20):1640-1642. doi: 10.1093/eurheartj/ehy777. No abstract available. PMID 30496563
- [Background] Caruso FR, Junior JC, Mendes RG, Sperling MP, Arakelian VM, Bassi D, Arena R, Borghi-Silva A. Hemodynamic and metabolic response during dynamic and resistance exercise in different intensities: a cross-sectional study on implications of intensity on safety and symptoms in patients with coronary disease. Am J Cardiovasc Dis. 2016 May 18;6(2):36-45. eCollection 2016. PMID 27335689
- [Background] Chow CK, Redfern J, Thiagalingam A, Jan S, Whittaker R, Hackett M, Graves N, Mooney J, Hillis GS. Design and rationale of the tobacco, exercise and diet messages (TEXT ME) trial of a text message-based intervention for ongoing prevention of cardiovascular disease in people with coronary disease: a randomised controlled trial protocol. BMJ Open. 2012 Jan 19;2(1):e000606. doi: 10.1136/bmjopen-2011-000606. Print 2012. PMID 22267690
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P. Microvascular coronary disease in women: role of the cardiopulmonary exercise testing. Int J Cardiol. 2013 Oct 3;168(3):3012-3. doi: 10.1016/j.ijcard.2013.04.055. Epub 2013 May 7. No abstract available. PMID 23664441
- [Derived] Li Y, Li C, Wen J, Cui M, Wei Q, Liu M, Chen Z, Fang H, Liu L, Fu J, Zhang J, Lyu S. Tai Chi as a mind-body exercise modulates endothelial function in coronary artery disease: A randomized clinical trial. Complement Ther Med. 2025 Sep;92:103201. doi: 10.1016/j.ctim.2025.103201. Epub 2025 Jun 18. PMID 40553955
- [Derived] Ma J, Zhang JW, Li H, Zhao LS, Guo AY, Chen ZH, Yuan W, Gao TM, Li YM, Li CH, Wang HW, Song B, Lu YL, Cui MZ, Wei QY, Lyu SJ, Yin HC. Safety and effectiveness of a Tai Chi-based cardiac rehabilitation programme for chronic coronary syndrom patients: study protocol for a randomised controlled trial. BMJ Open. 2020 Jul 5;10(7):e036061. doi: 10.1136/bmjopen-2019-036061. PMID 32624473
- See also: Wichita State University — http://www.researcherid.com/rid/C-4027-2012